CLINICAL TRIAL: NCT03354988
Title: Effect of Assisted Exercise on Musculoskeletal System and Growth in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, Associate Professor of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU 2015
Record Dates: First submitted 2016-03-19; First posted 2017-11-28 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Osteopenia Prematurity
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- physical exercise group (Active Comparator): For the exercise group, Intervention by doing physical exercise. systematic physical activity programs consisting of range-of-motion exercises with gentle compression, extension and flexion of all joints of both bilateral upper extremities; including the shoulder, elbow, and wrist and lower extremities; including the hip, knee and ankle, with a total of 12 joints. Each activity was about 10 min a day and was carried out 5 times per week for 4 weeks. This program was started after 1 week of birth. Physical activity continued until discharge from hospital.
  Interventions: Other: Physical exercise group
- Control group (Other): Other routine care activities such as bathing (every day) and kangaroo care (30 minutes/day), will be done for both the control
  Interventions: Other: Control group

INTERVENTIONS:
Other: Physical exercise group — For the exercise group, systematic physical activity programs consisting of range-of-motion exercises with gentle compression, extension and flexion of all joints of both bilateral upper extremities; including the shoulder, elbow, and wrist and lower extremities; including the hip, knee and ankle, with a total of 12 joints. Each activity was about 10 min a day and was carried out 5 times per week for 4 weeks. This program was started after 1 week of birth. Physical activity continued until discharge from hospital
  Arms: physical exercise group
Other: Control group — Other routine care activities such as bathing (every day) and kangaroo care (30 minutes/day), will be done for both the control
  Arms: Control group

SUMMARY:
The primary aim of this study is to assess whether physical activity programs in preterm infants improve bone mineralization as well as growth and reduce the risk of fractures.

The secondary aim is to include other potential benefits in terms of length of hospital stay, weaning from mechanical ventilation, feeding tolerance and adverse events

DETAILED DESCRIPTION:
This is a prospective randomized controlled clinical trial that will be conducted on 36 VLBW preterm infants admitted to the neonatal intensive care unit (NICU) - Ain Shams University

METHODS:

All the newborns included in the study will be subjected to the following:

1. Comprehensive history taking including:

   * Antenatal history: Maternal age, maternal diseases, maternal diabetic control, maternal infection (STORCH infection), maternal medication during this pregnancy, and last menstrual period.
   * Natal history: Gestational age, neonatal sex and mode of delivery.
   * Postnatal history: Respiratory distress and cyanosis.
   * Family history: Consanguinity, congenital anomalies, previous abortion, sibling death, and still birth.
2. Thorough clinical examination with particular emphasis on:

   * Assessment of Apgar scores at 1 and 5 minutes
   * Assessment of gestational age based on last menstrual period and confirmed by ultrasonography in early pregnancy if possible and Ballard scores
   * Complete examination including cardiac, chest, abdominal, and neurological examination.
3. Sample size calculation and Randomization:

   The sample size was calculated using power and sample size calculation program and was based on the previously reported intervention changes in Bone mineral density (BMD) following assisted exercise. A mean difference of 5.3 mg cm2 between the groups, with a standard deviation of 5.6 mg cm2 was used, based on the study by Considering a 0.05 significance level and power equal to 80%, an n of 19 patients per group was determined.

   Patients who will meet the inclusion criteria will be randomized into the physical exercise (n=18) and control (n=18) groups. Randomization will be made by birth order; the first born preterm infant will be recruited to the exercise group, the second to the control group, etc.
4. Standard neonatal care:

   * Babies admitted to NICU bathed, placed in incubator, attached to monitor.
   * Cannula inserted, IV fluids is started (Dexstrose10%) and IV antibiotics.
   * If there is respiratory distress: O2 or ventilation is started, usually feeds are delayed to day 2 or day 3 (or even later) according the severity of condition (clinical decision according to the attending neonatologist).
   * If no distress and the baby is well: trophic feeds is started (10ml/kg/day milk), feeds is increased in 10-20ml/kg/day according to baby tolerance, and the condition of the baby (clinical decision according to the attending neonatologist), IV fluids are reduced gradually.
5. Exercise protocol:

   The exercise protocol was designed for Infants in treatment and control groups received well defined interventions applied by the same trained occupational therapist, described as follows:

   For the exercise group, systematic physical activity programs consisting of range-of-motion exercises with gentle compression, extension and flexion of all joints of both bilateral upper extremities; including the shoulder, elbow, and wrist and lower extremities; including the hip, knee and ankle, with a total of 12 joints. Each activity was about 10 min a day and was carried out 5 times per week for 4 weeks. This program was started after 1 week of birth. Physical activity continued until discharge from hospital.

   Because tactile stimulation might have influenced growth and development, control subjects had a daily interactive period of holding and stroking but no range-of-motion activity. The time schedule of each activity was the same as the exercise group. Other routine care activities such as bathing (every day) and kangaroo care (30 minutes/day), will be done for both the control and exercise group subjects according to the neonatal intensive care unit (NICU) recommendations, however, without movement and standardized articular compression.
6. Laboratory investigation:

   * Complete blood count with differential leucocytic count.
   * Serum calcium concentration.
   * Serum phosphorous concentration.
   * Serum magnesium concentration.
   * Serum alkaline phosphates concentration.
   * Serum Alanine Aminotransferase (ALT).
   * Serum carboxy-terminal cross linked telopeptides of type 1 collagen (CTX).
   * Urinary calcium/phosphorous ratio.

   All the previous investigations will be done before at after the end of the exercise protocol for patients and control groups.
7. Bone mineralization will be assessed by measured by dual- energy x- ray absorptiometry (DEXA) :

   DEXA evaluates body composition (total body will be done after the end of the exercise protocol for patients and control groups by measuring:
   * Bone mineral Content (BMC, mg),
   * Bone Mineral Density (BMD, mg/ cm2),
   * Bone area (BA/ cm2),
   * Lean mass (LM, g) and
   * Fat mass (g).
8. Ethical Considerations:

Collected data will be used for study purpose only. The mothers of the newborns under study will be informed about the purpose of the study and the plan of work before agreeing to participate. They will be provided informed consent before the testing began. Study protocol will be presented to and approved by the Ethical Committee of the Scientific Research-Ain Shams University.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (gestational age <37 completed weeks) who did not receive physical therapy for any indication other than osteopenia of prematurity (e.g. severe contractures);
* Birth weight ≤ 1.500gm;
* Body size appropriate for gestational age;
* Postnatal age of ≥1 week with medically stable condition and favorable evolution that is presenting no associated diseases besides prematurity;
* Tolerating enteral feeds of either fortified breast milk or preterm formula at or above 100 kcal/kg/d.
* Not requiring oxygen or mechanical ventilation at the start of the exercise protocol.

Exclusion Criteria:

* Congenital or acquired anomaly of the Respiratory tract (i.e., diaphragmatic hernia, pulmonary hypoplasia, pulmonary sequestration, bronchogenic cysts);
* Other major congenital anomalies (congenital heart disease, neural tube defect, omphalocele, trisomy, etc.);
* Premature infants diagnosed with serious periventricular hemorrhaging (degrees 3 and 4) or serious sepsis;
* Use of medications (diuretics, methylxanthines and corticosteroids); Infants who had received major surgery within the first two weeks of life

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
serum calcium | 2 weeks
  mg/dL
serum PO4 | 2 weeks
  mg/dL
serum magnesium | 2 weeks
  mg/dL
ALP | 2 weeks
  IU/L
CTX | 2 weeks
  pg/mL
Whole body BMD | 2 weeks
  mg/cm2

CONTACTS AND LOCATIONS:
Overall Officials: rania elfarrash, assprofessor, Principal Investigator — Ain Shams univeristy
Locations (1):
- Ain shams university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No